CLINICAL TRIAL: NCT05145530
Title: Selective Nerve Root Block With Ultrasound Guidance Improves Surgical Outcome of Selective Discectomy in Patients With Multilevel Cervical Disc Disease: a Randomized Controlled Trial
Brief Title: Selective Nerve Root Block With Ultrasound Guidance Improves Surgical Outcome of Selective Discectomy in Patients With Multilevel Cervical Disc Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17300111
Record Dates: First submitted 2021-11-26; First posted 2021-12-06 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Selective Nerve Root Block; Selective Discectomy
MeSH Terms: interventions — Gene Fusion

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Active Comparator): selective anterior cervical discectomy and fusion (ACDF)
  Interventions: Procedure: selective anterior cervical discectomy and fusion (ACDF)
- Group SNRB (Experimental): US-guided selective nerve root block (SNRB) then selective anterior cervical discectomy and fusion (ACDF)
  Interventions: Procedure: SNRB+ selective anterior cervical discectomy and fusion (ACDF)

INTERVENTIONS:
Procedure: selective anterior cervical discectomy and fusion (ACDF) — selective anterior cervical discectomy and fusion (ACDF)
  Arms: Group C
Procedure: SNRB+ selective anterior cervical discectomy and fusion (ACDF) — US-guided selective nerve root block (SNRB) + selective anterior cervical discectomy and fusion (ACDF)
  Arms: Group SNRB

SUMMARY:
Disc degeneration is a natural part of growing older. Up to 60% of asymptomatic people have MRI findings that are positive. As a result, MRI only provides morphological information and may not be able to determine the clinical significance of the findings.

DETAILED DESCRIPTION:
Many authors believe that patients who suffer from cervical radiculopathy as a result of degenerative disease and have multilevel pathology on imaging studies still have moderate surgical outcomes. This occurs due to a misdiagnosis or the need to perform surgery on multiple levels despite a single painful lesion.

Although the complication rate for 1- and 2-level ACDF is so low that it is considered one of the safest procedures in spine surgery. There is concern that increasing levels of fusion will lead to more complications, such as a higher incidence of persistent axial neck pain, dysphagia, and vertebral artery injury, as well as more postoperative pain and higher narcotic dosages.

ELIGIBILITY:
Inclusion Criteria:

* all patients presented with unilateral brachialgia due to multilevel cervical disc disease

Exclusion Criteria:

* multilevel cervical disc disease who had bilateral brachialgia,
* myelopathy, double crush syndrome,
* ossified posterior longitudinal ligament (OPLL),
* combined anterior and posterior pathology requiring posterior decompression

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
pain intensity | 24 hours postoperative
  Visual analogue score (VAS): 0= no pain, 10= worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kreitz TM, Hollern DA, Padegimas EM, Schroeder GD, Kepler CK, Vaccaro AR, Hilibrand AS. Clinical Outcomes After Four-Level Anterior Cervical Discectomy and Fusion. Global Spine J. 2018 Dec;8(8):776-783. doi: 10.1177/2192568218770763. Epub 2018 Apr 24. PMID 30560028
- [Background] McClure JJ, Desai BD, Shabo LM, Buell TJ, Yen CP, Smith JS, Shaffrey CI, Shaffrey ME, Buchholz AL. A single-center retrospective analysis of 3- or 4-level anterior cervical discectomy and fusion: surgical outcomes in 66 patients. J Neurosurg Spine. 2020 Oct 9;34(1):45-51. doi: 10.3171/2020.6.SPINE20171. Print 2021 Jan 1. PMID 33036003
- [Background] Ross DA, Ross MN. Diagnosis and Treatment of C4 Radiculopathy. Spine (Phila Pa 1976). 2016 Dec 1;41(23):1790-1794. doi: 10.1097/BRS.0000000000001620. PMID 27054454